CLINICAL TRIAL: NCT03188978
Title: High-intensity Atorvastatin for Arteriovenous Fistula Failure (HAFF): A Feasibility Pilot Study
Acronym: HAFF
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Unable to recruit
Sponsor: Albany Medical College (Other)
Responsible Party: Principal Investigator, Loay Salman, MD, Professor of Medicine, Albany Medical College
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HAFF
Record Dates: First submitted 2017-06-12; First posted 2017-06-16 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Primary Arteriovenous Fistula Failure
MeSH Terms: interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment (Experimental): Atorvastatin 40mg once daily orally for 8 weeks starting 2 weeks before AVF creation
  Interventions: Drug: Atorvastatin 40mg
- Placebo (Placebo Comparator): 1 tablet once daily orally for 8 weeks starting 2 weeks before AVF creation
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Atorvastatin 40mg — one 40mg tablet daily for 8 weeks starting 2 weeks before the AVF creation.
  Other Names: Lipitor 40mg tablets
  Arms: Treatment
Other: Placebo — one tablet daily for 8 weeks starting 2 weeks before the AVF creation.
  Arms: Placebo

SUMMARY:
Primary failure is the most common complication of newly created arteriovenous fistulas (AVFs) and an important contributor to end stage renal disease (ESRD) patients' morbidity and mortality. Recently, the investigators have found that high intensity atorvastatin (40 mg/day) reduces AVF primary failure significantly when compared to other statins or no statin treatment in three separate prospective and retrospective studies done in collaboration with the University of Miami. Based on these findings and considering the necessity for a therapy to improve AVF maturation rates, the investigators propose the realization of a feasibility pilot double blinded randomized controlled trial (RCT). In this study, a total of 50 patients will be randomly allocated to receive high intensity atorvastatin (40 mg daily) or placebo starting at two weeks before surgery and until the end of the observational period (6 weeks after surgery). Present trial will reveal crucial feasibility information such as the appropriateness of the eligibility criteria, patient recruitment and retention rates, compliance, adverse events, efficacy of patient follow-ups, and readiness of the facilities and involved personnel; while having as a secondary endpoint the predictive measurements of diameter and AVF blood flow 6 weeks after fistula creation useful for the estimation of the probable effect of proposed intervention. Here, the investigators aim to pave the way for a future multicenter Phase II RCT seeking to prove the efficacy of atorvastatin therapy as a perioperative intervention to reduce AVF primary failure.

DETAILED DESCRIPTION:
STUDY BACKGROUND AND PURPOSE. Approximately, 30-50% of newly created arteriovenous fistulas (AVF) never mature independently to support hemodialysis, leading to salvage interventions or abandonment of the fistula and creation of a new dialysis access. Failed AVFs are thus associated with increased morbidity, mortality and health care expenditures.

Only two published studies have assessed the effect of statins on AVF primary failure, with contrasting results. Pisoni et al. concluded that statins did not improve AVF maturation, using a retrospective analysis of 317 patients and pooling all statins together as a drug class. Unfortunately, this approach overlooks the potential pleiotropic effects of distinct drugs on AVF remodeling. Overcoming the limitations of Pisoni et al.'s study, the investigators recently published a manuscript evaluating the benefits of three different statins (atorvastatin, rosuvastatin and simvastatin) on AVF outcomes using a retrospective analysis of 535 patients. In this work done in collaboration with the University of Miami, the investigators found a highly statistical significant risk reduction (76%, odds ratio [OR] 0.18, p=0.005) of AVF primary failure by atorvastatin. No other statins significantly improved AVF maturation in this cohort. Interestingly, this study showed that atorvastatin is particularly beneficial for one-stage AVF (96% risk reduction, OR 0.03, p=0.005) and, that higher doses of the drug are associated with lower rates of primary failure in one-stage fistulas. Two more studies done by the same group, a prospective and another retrospective, also support this finding indicating that the use of statins prior to fistula creation is beneficial for the unassisted survival of the AVF.

Compared to other statins, atorvastatin has a distinctive physicochemical and pharmacokinetic profile. These characteristics could explain the differential pleiotropic action of atorvastatin in investigators' study, and why it is superior to its counterparts in improving vascular remodeling after AVF creation.

Based on above findings, the investigators propose a pilot clinical trial to evaluate the feasibility of a study involving ESRD patients undergoing AVF surgery at AMC. Indeed, the investigators long-term goal is the realization of a large multicenter Phase II Randomized Controlled Trial (RCT) to test the efficacy of atorvastatin as a safe and inexpensive therapeutic intervention for the reduction of AVF primary failure.

The present proposal will be implemented as presented in the following specific aim (SA): Evaluate the feasibility of performing a RCT with patients taking atorvastatin and undergoing AVF surgery at Albany Medical College.

The primary outcome in this study will be our ability to recruit the patients and follow them up after surgery for 6 weeks through the standard clinical and laboratory tests for ESRD patients undergoing this procedure. This pilot study will help evaluate important feasibility aspects such as the appropriateness of the eligibility criteria, patient recruitment and retention rates, compliance, competency of personnel and site (which include availability and readiness of facilities and study coordinators, pharmacists, nurses, and others) and also to document any adverse event.

The secondary endpoints will be the ultrasonographic (US) measurements of diameter and AVF blood flow 6 weeks after fistula creation. Diameter and blood flow at 6-week have been shown to be of value as predictors of AVF maturation, and having this information is useful to better assess the sample size for future main trials after obtaining the variance estimation of proposed intervention. This information will help to cut study time and expenses in the future.

STUDY DESIGN Enrollment. Patients scheduled to undergo AVF creation will be evaluated by participating surgeons at Albany Medical College approximately one month prior to surgery. Pre-operative vascular assessment will be performed by Doppler ultrasound and the patient's chart will be reviewed for additional relevant information pertinent to the surgery or the proposed intervention. Potential candidates will be approached by the PI and/or vascular surgeons, and clinical research coordinator (CRC) to enroll in this study. If subject agrees the informed consent is obtained, blood will be collected for a baseline Liver test function (LFT), C-reactive protein (CRP), creatine phosphokinase (CPK), and lipid profile, and the patient's clinical information will be entered into Qualtrics (clinical research management software). If the results of the baseline blood panel do not warrant an exclusion, and eligibility criteria are met, patients will be contacted and they will receive the study medication and date they should start the therapy (2 weeks prior to surgery). The patient's primary doctor will be notified and a note will be entered into the patient's electronic record to inform of his/her participation in the study. The day prior to treatment initiation, patients will be called as a reminder. Investigators' goal is to enroll fifty patients, who will be randomized to receive either atorvastatin (40mg, once daily) or placebo. The active drug and matching placebo will be compounded by Pfizer Inc. (New York, NY), the original producer and owner of Lipitor. To ensure that results will not be biased, neither the participants nor the researchers will know which patient belong to the placebo group, nor the statin group. Each patient will participate in the study for eight weeks. This study will be completed in no more than 2 years.

INFORMED CONSENT (ICF). The investigators will follow the AMC Institutional Review Board and U.S. Department of Health & Office for Human Research protection guidelines. Subjects will be recruited for this study from the hemodialysis and chronic kidney disease populations at Albany Medical College. All patients will receive the same standard of care independently of their enrollment, compliance or retention in the study. Subjects will be free to withdraw from the study at will.

SAMPLE SIZE and STATISTICAL considerations. This feasibility pilot trial is focused at site and investigator level and it is not required to provide power calculation. However, this study must be seen in the context of the future Phase II trial that should result from it, as pilot trial size can impact the overall sample size across both the main and pilot trials combined. The trial sample size of 25 patients per arm (50 patients in total) was selected according Whitehead et al., and it could give investigators the additional advantage of calculating the standardized variance of our secondary endpoints if a medium experimental effect size is observed.

FOLLOW-UP. Follow-up of patients will be performed by the PI as well as the CRC. The day of the AVF surgery, patients will be interviewed to assess compliance and adverse events. If a patient reports significant side effects, she/he will be asked to discontinue the therapy and the final blood panel will be ordered (LFT, CRP, CPK, and lipids). Otherwise, patients will be reminded to continue with the treatment until their next follow-up appointment with the vascular surgeon 2-3 weeks after operation (5-6 weeks after treatment initiation); when a LFT will be done following the American College of Cardiologists/American Heart Association (ACC/AHA) guidelines for monitoring patients who have begun statin therapy. If any surgical complications arise prior to the final evaluation, these will be recorded and treated accordingly, and the study treatment will be discontinued. The day of the final evaluation (8 weeks after intervention initiation), compliance will be evaluated as well as the AVF status will be assessed by Doppler ultrasound and auscultation; the secondary endpoints will be recorded (AVF diameter and blood flow) and a final lab panel will be drawn as done at baseline. Additional outcomes will include changes in lipid profiles, LFTs, and CRP from baseline; frequency of adverse effects; as well as patient compliance and retention rates in each arm of the study.

SUBJECT POPULATION. Investigators will enroll fifty subjects aged over 18 years old with stage 4 or 5 CKD scheduled to undergo AVF creation from the clinic at Albany Medical College. AMC has a long history of providing medical care to underrepresented minorities. In investigators' previous studies women composed 45% of the study population, 30% were black, 10% were Hispanic, and 5% other minority races (Asian, Native American, etc.). Investigators anticipate similar rates of inclusion of women and minorities in the current proposal. It has been reported an increased AVF maturation rate failure in women, therefore, they could potentially benefit more from the proposed intervention. Overall, investigators are not aiming at recruiting patients from specific ethnic or racial group in this study.

DATA ANALYSIS. Analyses will be performed after all patients have completed the study by the participating biostatistician, the PI or other study researchers under their supervision. In addition to the baseline and follow-up laboratory tests, relevant clinical information will be collected from patients including age, gender, ethnicity, prior vascular access and surgical history, concurrent medications, and comorbidities. With the exception of numerical variables such as laboratory values and age, all other clinical variables will be annotated as binary. At the conclusion of the study, the patient characteristics of both treatment arms will be compared to assure their equivalency. The study data will be analyzed following the recommended intention-to-treat protocol, in which all enrolled patients are accounted for at the end of the observational period. If differences in baseline characteristics are not statistically significant (p<0.05), a Fisher's exact test will be used to compare AVF blood flow and diameter between study arms. On the other hand, if significant differences are detected in one or more relevant baseline variables, logistic regression analyses will be used to adjust for the effect of baseline covariables on the secondary endpoints. An evaluation of compliance, retention rates and adverse effects will be also performed for all the patients and the distinct subpopulations. If compliance is found to be an issue, the analysis of endpoints using a per-protocol approach will be considered. The SAS statistical software package, version 9.2 (Cary, NC), will be used for all statistical analyses.

RISKS. Atorvastatin has a well-established safety and adverse reactions profiles and is already used in the hemodialysis population for different indications. Chronic Kidney Disease participants enrolled in this trial have elevated risks of cardiovascular events, and although only statin-naïve patients or statin-free in the last 6 months prior to enrollment will be eligible to participate, it is likely that many of these patients already have an indication for statin treatment. In order to minimize the occurrence of potential adverse effects, the investigators will carefully evaluate the potential candidates for the study prior to the enrollment and will follow the 2013 ACC/AHA blood cholesterol guidelines recommendations. The investigators will do fasting lipid panel, hepatic transaminase levels, CRP and CPK at baseline, at 5-6 weeks after therapy initiation, and at the final follow up at 8 weeks of therapy. There are no additional risks associated with the procedures that are going to be performed in this study other than phlebotomy and surgery-related complications.

BENEFITS. The great potential benefit of Atorvastatin in this study is to reduce primary AVF failure in the treated group. Knowledge obtained from this pilot study will be of paramount importance and may lead to a phase II trial that will pave the way toward an effective treatment of AVF primary failure with a widely available medication.

ELIGIBILITY:
Inclusion Criteria:

* age>18 years of age;
* stage 4 or 5 CKD;
* one-stage AVF surgery is planned (radiocephalic or brachiocephalic);
* and statin-naïve or at least 6 months from last statin use.

Exclusion Criteria:

* revision of an existing AVF instead of a de novo access;
* known intolerance or hypersensitivity to statins;
* active liver disease;
* elevation in AST, ALT or CPK of more than 3 times the upper limit of normal;
* baseline LDL<40 mg/dL;
* coadministration of strong interacting drugs;
* any condition in which statins are contraindicated;
* involvement in another trial where the intervention may confound the outcome of this trial.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Patient recruitment rate (in percent) | 104 weeks
  The patient recruitment rate (in percent) is an important parameter to evaluate the feasibility of the study and to plan future Phase II trials.
Patient retention rate (in percent) | 104 weeks
  The patient retention rate (in percent) is an important parameter to evaluate the feasibility of the study and to plan future Phase II trials.
Patient compliance (in percent) | 104 weeks
  The patient compliance (in percent) is an important parameter to evaluate the feasibility of the study and to plan future Phase II trials.
Rate of adverse events (in percent) | 104 weeks
  The rate of adverse events (in percent) is an important parameter to evaluate the safety of the study and it is important to plan future Phase II trials.

SECONDARY OUTCOMES:
Ultrasonographic measurement of AVF blood flow (in milliliter per minute). | 104 weeks
  The predictive measurement of AVF blood flow (in milliliter per minute) 6 weeks after fistula creation is useful for the estimation of the probable effect of proposed intervention in order to better assess the sample size for subsequent RCT.
Ultrasonographic measurements of diameter (in millimeters). | 104 weeks
  The predictive measurements of diameter (in millimeters) 6 weeks after fistula creation is useful for the estimation of the probable effect of proposed intervention in order to better assess the sample size for subsequent RCT.

CONTACTS AND LOCATIONS:
Overall Officials: Loay Salman, MD,MBA, Principal Investigator — Albany Medical College
Locations (1):
- Albany Medical College, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: No
No personal data will be transfer outside AMC. Study paper records, computer files, and communications will be appropriately safeguarded by study personnel and the IT department from unauthorized access. Name or any other data that might identify patients will not be used in any reports or publications resulting from this study. Password-protected computers will be utilized, and the identity of subjects will be maintained separately from computerized data forms. Only the primary investigator and members of the research team who contact the subjects will have access to collected information in a need to know basis. All clinical data and biological specimens obtained will be linked to the individual subject by only a unique study identification code (master-key). The PI will keep the master-key secure and confidential in his office, and only he and the CRC will have access to the master-key.

REFERENCES:
- [Background] Huijbregts HJ, Bots ML, Wittens CH, Schrama YC, Moll FL, Blankestijn PJ; CIMINO study group. Hemodialysis arteriovenous fistula patency revisited: results of a prospective, multicenter initiative. Clin J Am Soc Nephrol. 2008 May;3(3):714-9. doi: 10.2215/CJN.02950707. Epub 2008 Feb 6. PMID 18256379
- [Background] Schinstock CA, Albright RC, Williams AW, Dillon JJ, Bergstralh EJ, Jenson BM, McCarthy JT, Nath KA. Outcomes of arteriovenous fistula creation after the Fistula First Initiative. Clin J Am Soc Nephrol. 2011 Aug;6(8):1996-2002. doi: 10.2215/CJN.11251210. Epub 2011 Jul 7. PMID 21737851
- [Background] Bashar K, Zafar A, Elsheikh S, Healy DA, Clarke-Moloney M, Casserly L, Burke PE, Kavanagh EG, Walsh SR. Predictive parameters of arteriovenous fistula functional maturation in a population of patients with end-stage renal disease. PLoS One. 2015 Mar 13;10(3):e0119958. doi: 10.1371/journal.pone.0119958. eCollection 2015. PMID 25768440
- [Background] Pisoni R, Barker-Finkel J, Allo M. Statin therapy is not associated with improved vascular access outcomes. Clin J Am Soc Nephrol. 2010 Aug;5(8):1447-50. doi: 10.2215/CJN.02740310. Epub 2010 May 27. PMID 20507962
- [Background] Martinez L, Duque JC, Escobar LA, Tabbara M, Asif A, Fayad F, Vazquez-Padron RI, Salman LH. Distinct impact of three different statins on arteriovenous fistula outcomes: a retrospective analysis. J Vasc Access. 2016 Nov 2;17(6):471-476. doi: 10.5301/jva.5000612. Epub 2016 Oct 15. PMID 27768209
- [Background] Robbin ML, Greene T, Cheung AK, Allon M, Berceli SA, Kaufman JS, Allen M, Imrey PB, Radeva MK, Shiu YT, Umphrey HR, Young CJ; Hemodialysis Fistula Maturation Study Group. Arteriovenous Fistula Development in the First 6 Weeks after Creation. Radiology. 2016 May;279(2):620-9. doi: 10.1148/radiol.2015150385. Epub 2015 Dec 22. PMID 26694050
- [Background] Whitehead AL, Julious SA, Cooper CL, Campbell MJ. Estimating the sample size for a pilot randomised trial to minimise the overall trial sample size for the external pilot and main trial for a continuous outcome variable. Stat Methods Med Res. 2016 Jun;25(3):1057-73. doi: 10.1177/0962280215588241. Epub 2015 Jun 19. PMID 26092476
- [Background] Teare MD, Dimairo M, Shephard N, Hayman A, Whitehead A, Walters SJ. Sample size requirements to estimate key design parameters from external pilot randomised controlled trials: a simulation study. Trials. 2014 Jul 3;15:264. doi: 10.1186/1745-6215-15-264. PMID 24993581
- [Background] Liao JK, Laufs U. Pleiotropic effects of statins. Annu Rev Pharmacol Toxicol. 2005;45:89-118. doi: 10.1146/annurev.pharmtox.45.120403.095748. PMID 15822172
- [Background] Bonetti PO, Lerman LO, Napoli C, Lerman A. Statin effects beyond lipid lowering--are they clinically relevant? Eur Heart J. 2003 Feb;24(3):225-48. doi: 10.1016/s0195-668x(02)00419-0. No abstract available. PMID 12590901
- [Background] Schachter M. Chemical, pharmacokinetic and pharmacodynamic properties of statins: an update. Fundam Clin Pharmacol. 2005 Feb;19(1):117-25. doi: 10.1111/j.1472-8206.2004.00299.x. PMID 15660968
- [Background] Mason RP. Molecular basis of differences among statins and a comparison with antioxidant vitamins. Am J Cardiol. 2006 Dec 4;98(11A):34P-41P. doi: 10.1016/j.amjcard.2006.09.018. Epub 2006 Oct 10. PMID 17126678
- [Background] Tabbara M, Duque JC, Martinez L, Escobar LA, Wu W, Pan Y, Fernandez N, Velazquez OC, Jaimes EA, Salman LH, Vazquez-Padron RI. Pre-existing and Postoperative Intimal Hyperplasia and Arteriovenous Fistula Outcomes. Am J Kidney Dis. 2016 Sep;68(3):455-64. doi: 10.1053/j.ajkd.2016.02.044. Epub 2016 Mar 22. PMID 27012909
- [Background] Duque JC, Martinez L, Tabbara M, Dvorquez D, Mehandru SK, Asif A, Vazquez-Padron RI, Salman LH. Arteriovenous fistula maturation in patients with permanent access created prior to or after hemodialysis initiation. J Vasc Access. 2017 May 15;18(3):185-191. doi: 10.5301/jva.5000662. Epub 2017 Feb 15. PMID 28218361
- [Background] Stone NJ, Robinson JG, Lichtenstein AH, Bairey Merz CN, Blum CB, Eckel RH, Goldberg AC, Gordon D, Levy D, Lloyd-Jones DM, McBride P, Schwartz JS, Shero ST, Smith SC Jr, Watson K, Wilson PW, Eddleman KM, Jarrett NM, LaBresh K, Nevo L, Wnek J, Anderson JL, Halperin JL, Albert NM, Bozkurt B, Brindis RG, Curtis LH, DeMets D, Hochman JS, Kovacs RJ, Ohman EM, Pressler SJ, Sellke FW, Shen WK, Smith SC Jr, Tomaselli GF; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2013 ACC/AHA guideline on the treatment of blood cholesterol to reduce atherosclerotic cardiovascular risk in adults: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. Circulation. 2014 Jun 24;129(25 Suppl 2):S1-45. doi: 10.1161/01.cir.0000437738.63853.7a. Epub 2013 Nov 12. No abstract available. PMID 24222016
- [Background] Foundation NK. KDOQI clinical practice guidelines and clinical practice recommendations for 2006 updates: hemodialysis adequacy, peritoneal dialysis adequacy and vascular access. Am J Kidney Dis. 2006;48(Suppl 1):S1-S322.
- [Background] Dember LM, Imrey PB, Beck GJ, Cheung AK, Himmelfarb J, Huber TS, Kusek JW, Roy-Chaudhury P, Vazquez MA, Alpers CE, Robbin ML, Vita JA, Greene T, Gassman JJ, Feldman HI; Hemodialysis Fistula Maturation Study Group. Objectives and design of the hemodialysis fistula maturation study. Am J Kidney Dis. 2014 Jan;63(1):104-12. doi: 10.1053/j.ajkd.2013.06.024. Epub 2013 Aug 28. PMID 23992885
- [Background] Gupta SK. Intention-to-treat concept: A review. Perspect Clin Res. 2011 Jul;2(3):109-12. doi: 10.4103/2229-3485.83221. PMID 21897887
- [Background] Robbin ML, Chamberlain NE, Lockhart ME, Gallichio MH, Young CJ, Deierhoi MH, Allon M. Hemodialysis arteriovenous fistula maturity: US evaluation. Radiology. 2002 Oct;225(1):59-64. doi: 10.1148/radiol.2251011367. PMID 12354984